CLINICAL TRIAL: NCT04403620
Title: HYPORT: A Phase I/II Study of Hypofractionated Post-operative Radiation Therapy for Head and Neck Squamous Cell Carcinoma
Brief Title: HYPORT: A Phase I/II Study of Hypofractionated Post-operative Radiation Therapy for Head and Neck Cancer
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Dominic Moon, Assistant Professor, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: STU 2020-0522
Record Dates: First submitted 2020-05-14; First posted 2020-05-27 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Squamous Cell Carcinoma of Head and Neck
Keywords: Radiation Dose Hypofractionation; Adjuvant Radiotherapy
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Intervention Model Description: Dose/fractionation finding Phase 1 study, followed by a randomized Phase 2 study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Conventionally fractionated radiotherapy (Active Comparator): 60 Gy in 30 fractions, 5 fractions/week
  Interventions: Radiation: Intensity-modulated Radiation Therapy (IMRT)
- Hypofractionated radiotherapy (Experimental): Dose and fractionation determined by Phase I:
  Level 1: 44.4 Gy in 12 fractions, 4 fractions/week
  Level 0: 46.5 Gy in 15 fractions, 5 fractions/week
  Level -1: 52 Gy in 20 fractions, 5 fractions/week
  Level -2: 50 Gy in 20 fractions, 5 fractions/week
  Interventions: Radiation: Intensity-modulated Radiation Therapy (IMRT)

INTERVENTIONS:
Radiation: Intensity-modulated Radiation Therapy (IMRT) — Patients will receive adjuvant radiation therapy using intensity-modulated radiation therapy (IMRT) within 8 weeks of surgical resection

SUMMARY:
There is a strong radiobiological and economic rationale for hypofractionated radiation therapy in head and neck cancer. Phase 1 of the trial aims to assess the acute toxicity and tolerability of hypofractionated radiation therapy in the post-operative setting, and to determine the dose/fractionation for Phase 2. Phase 2 aims to establish non-inferiority of swallowing-related quality of life and to assess the toxicity and efficacy of hypofractionated radiation therapy compared to conventionally fractionated radiation therapy in the post-operative setting.

DETAILED DESCRIPTION:
The trial will assess the effects of aggressive hypofractionated radiation therapy in patients with oral cavity, oropharynx, hypopharynx, or larynx cancer after surgical resection with pathology showing intermediate risk factors requiring post-operative radiation therapy without concurrent chemotherapy. During Phase 1, the maximum tolerated dose/fractionation and tolerability will be determined. During Phase 2, patients will be randomized between conventionally fractionated radiation therapy (6 weeks) vs. hypofractionated radiation therapy (3 weeks) to establish non-inferiority of hypofractionated radiation therapy.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria will be the same for Phase I and Phase II.

1. Pathologically proven diagnosis of stage I-IVB squamous cell carcinoma of the oral cavity, oropharynx, hypopharynx, or larynx status post gross total resection with pathology showing one or more of the following intermediate risk factors:

   * T3/4 disease (AJCC 8th edition), positive lymph node(s), close margin(s), perineural invasion, and/or lymphovascular invasion
   * Close margin(s) defined as either:

     * Final patient margin of <5 mm without disease on ink OR
     * Initial positive margin in the specimen regardless of the final patient margin (e.g. if resection margin on the initial specimen is positive, final patient margin after subsequent resections can be ≥5 mm and still be considered close margin)
2. Age ≥18 years
3. ECOG performance status 0-2
4. Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and for 90 days following completion of therapy.

   Medically acceptable birth control (contraceptives) includes:
   * approved hormonal contraceptives (such as birth control pills, patch or ring; Depo-Provera, Implanon), or
   * barrier methods (such as condom or diaphragm) used with a spermicide

   Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.

   A female of child-bearing potential is any woman (regardless of sexual orientation, having undergone a tubal ligation, or remaining celibate by choice) who meets the following criteria:
   * Has not undergone a hysterectomy or bilateral oophorectomy; or
   * Has not been naturally postmenopausal for at least 12 consecutive months (i.e., has had menses at any time in the preceding 12 consecutive months).
5. Negative serum or urine pregnancy test within 2 weeks before registration for women of childbearing potential.
6. Ability to understand and the willingness to sign a written informed consent

Exclusion Criteria:

Phase I:

1. Distant metastasis
2. Stage I and II glottic squamous cell carcinoma
3. High risk factors following surgical resection requiring concurrent chemotherapy: final positive margin(s) and/or extranodal extension
4. Feeding tube dependence at baseline assessment.
5. Synchronous non-skin cancer primaries outside of the oropharynx, oral cavity, larynx, and hypopharynx except for low- and intermediate-risk prostate cancer and synchronous well-differentiated thyroid cancer. For prostate cancer, patient should not be receiving active treatment. For thyroid cancer, thyroid surgery may occur before or after treatment, provided all other eligibility criteria are met.
6. Prior invasive malignancy with an expected disease-free interval of less than 3 years
7. Prior radiotherapy to the region of the study cancer that would result in overlap of radiation fields
8. Subjects may not be receiving any other investigational agents for the treatment of the cancer under study.
9. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that, in the opinion of the investigator, would limit compliance with study requirements
10. Subjects must not be pregnant or nursing due to the potential for congenital abnormalities and the potential of this regimen to harm nursing infants.
11. History of severe immunosuppression, including HIV, and organ or autologous or allogeneic stem cell transplant

Phase II:

The exclusion criteria will be the same as Phase I except for feeding tube dependence. Patients who are feeding tube dependent are excluded from Phase I to accurately assess treatment associated toxicity affecting swallowing and oral intake. During Phase II, patients who are feeding tube dependent will be eligible to enroll and stratified at randomization.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2020-07-28 (Actual); Primary Completion 2027-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Phase 1: Maximally tolerated dose of hypofractionated radiation therapy | 3 months
  Dose and fractionation to be used for Phase 2
Phase 2: Swallowing-related patient-reported quality of life | 12 months
  MD Anderson Dysphagia Inventory (MDADI) composite score: 20-100, higher scores mean better quality of life

SECONDARY OUTCOMES:
Clinician-reported acute toxicities | 1-3 months
  CTCAE v5.0
Clinician-reported late toxicities | 6-24 months
  CTCAE v5.0
Locoregional control | 12-24 months
Progression free survival | 12-24 months
Swallowing-related patient-reported quality of life | 1-24 months
  MD Anderson Dysphagia Inventory (MDADI): 20-100, higher scores mean better quality of life
Head and neck patient-reported quality of life | 1-24 months
  University of Washington QOL questionnaire (UW-QOL): 0-100, higher scores mean better quality of life
Xerostomia-related patient-reported quality of life | 1-24 months
  University of Michigan Xerostomia questionnaire (XQ): 0-100, higher scores mean worse quality of life
General patient-reported quality of life | 1-24 months
  EuroQol-5 dimensions (EQ-5D-5L): 1-5, higher scores mean worse quality of life
Feeding tube dependence | 1-24 months
  Feeding tube dependence defined as daily use of the feeding tube with ≥2 nutritional supplements (e.g. Ensure, Boost, etc.) per day at the time of enrollment on trial

CONTACTS AND LOCATIONS:
Overall Officials: Dominic Moon, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- University of Texas Southwestern Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No